CLINICAL TRIAL: NCT01019252
Title: Compensatory Executive Functioning Skills Training in Adolescents With ADHD
Brief Title: Skills Training for Adolescents With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Steven A. Safren, Director, Behavioral Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH083063 (NIH); R34MH083063 (NIH); DDTR B4-TBI (Other Grant/Funding Number: National Institute of Mental Health)
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Adolescent; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT for ADHD first, then follow-up (Experimental): Participants received Cognitive Behavioral Therapy following randomization.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Wait list first, then CBT for ADHD (No Intervention): Cross-over: Participants were assigned to a wait list after the initial assessment. They received Cognitive Behavioral Therapy after the 4 month assessment.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Participants are provided with education about ADHD and instruction in organizational skills, reducing distractibility, and adaptive thinking.
  Other Names: Compensatory executive skills training
  Arms: CBT for ADHD first, then follow-up

SUMMARY:
The proposed study will be an initial test of a cognitive-behavioral intervention for adolescents with ADHD who are receiving medication treatment. It is based on our successful work with adults with ADHD who have been treated with medicines but are still having symptoms. It involves learning skills for organization and planning, attention, and mood.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is a prevalent, distressing, and interfering condition that affects between 2% and 6% of adolescents. Although medications have been widely used as an effective treatment for many years as the sole treatment for ADHD, for many, clinically significant and interfering continued symptoms remain. Even after medication treatment, adolescents still experience residual ADHD symptoms and continue to have problems with inattention, concentration, disorganization, and other symptoms. However, research suggests that adolescents who have received some benefit from medication treatment can then experience further symptom reduction from participation in skills-based cognitive behavioral therapy. This study, adapted from a similar research study for adults with ADHD, will examine whether cognitive behavioral therapy (CBT) plus medication is more effective at treating ADHD than medication therapy alone in adolescents with ADHD.

Eligible participants will be randomly assigned to receive twelve weekly treatment sessions either immediately upon enrolling in the study or after a four-month waiting period. Questionnaires (that participants complete and ones that are done with an interviewer) will be used to assess participants' ADHD symptoms at study entry, after receiving the treatment, and at 4 month follow-up. Parents will have some involvement in therapy.

Note: participants must be able to come to Boston or another study location in the Greater Boston area for 4 assessment visits and 12 weekly therapy visits in order for participation to be feasible.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 14 and 18
* In high school
* Principal Diagnosis of ADHD
* Stable prescription of Medications for ADHD
* ADHD has childhood onset
* Clinically significant ADHD symptoms

Exclusion Criteria:

* Organic Mental Disorders
* Active Substance Abuse or Dependence
* Diagnosis of Conduct Disorder
* Mental Retardation or Pervasive Developmental Disorder
* Active Suicidality
* Previous History of CBT Therapy in adolescence
* Other condition interfering with consent or participation

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2009-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Safren, Ph.D., Principal Investigator — University of Miami; Susan E Sprich, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Sprich SE, Safren SA, Finkelstein D, Remmert JE, Hammerness P. A randomized controlled trial of cognitive behavioral therapy for ADHD in medication-treated adolescents. J Child Psychol Psychiatry. 2016 Nov;57(11):1218-1226. doi: 10.1111/jcpp.12549. Epub 2016 Mar 17. PMID 26990084

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through passive methods (e.g., local radio advertising, flyers, social media), active outreach (e.g., mailing through the Research Patient Data Registry), and physician referrals.
Pre-assignment Details: 66 adolescents completed baseline eligibility procedures. 2 opted-out of treatment due to logistical constraints.18 were excluded pre-randomization: 6 exclusionary psychiatric comorbidity, 5 clinician-rated severity below threshold, for 4 ADHD not primary diagnosis, and 2 not taking ADHD medication, 1 had a medical condition that would interfere.
Groups:
- CBT for ADHD First, Then Follow-up: All participants completed seven modules of treatment over twelve sessions, ten of which were 1:1 with the therapist and adolescent, and two of which also included the parent. Two additional optional parent-only sessions were offered as well. For each 1:1 session the parent was included for approximately ten minutes, generally at the end of the session, to discuss progress, the course of intervention content, and how the parent could assist with any take-home practice. 21 of the participants crossed-over to the wait list condition (received no further treatment) between the 4-month and 8-month assessments.
  Modules were adapted from the PI's intervention designed for ADHD in adults. Modules included: psychoeducation and organization/planning (4 session); distractibility (2 sessions); adaptive thinking/cognitive restructuring (2 sessions); procrastination (1 session); parent-adolescent sessions (2 sessions); parent-only sessions (1 session); relapse prevention (1 session).
- Wait List First, Then CBT for ADHD: Participants initially assigned to the wait list were informed by the research assistant that they had been randomized to the wait list condition. For those who were still willing to cross-over to receive CBT, the research assistant contacted parents to schedule the 4-month assessment visit with the independent evaluator and the first CBT session after the evaluation for participants. 19 participants crossed-over to receive CBT between the 4-month and 8-month assessments. Of the 19 who crossed-over, 15 completed the CBT treatment.
Period: Initial CBT for ADHD vs. Wait List
Arm/Group | CBT for ADHD First, Then Follow-up | Wait List First, Then CBT for ADHD
Started | 24 (Stratified based on biological sex and clinician-rated severity (CGI score)) | 22 (Stratified based on biological sex and clinician-rated severity (CGI score))
Completed | 21 | 22
Not Completed | 3 | 0
Not completed — Time constraints | 2 | 0
Not completed — Moved out of Boston area | 1 | 0
Period: Wait List Cross-over to CBT for ADHD
Arm/Group | CBT for ADHD First, Then Follow-up | Wait List First, Then CBT for ADHD
Started | 21 (Lost to follow up, did not start treatment following wait list completion (n=3)) | 22
Completed | 21 | 15
Not Completed | 0 | 7
Not completed — Time constraints | 0 | 2
Not completed — Lost to Follow-up | 0 | 5

BASELINE CHARACTERISTICS:
Population: Intention to treat analysis (ITT)
Groups:
- CBT First, Then Follow-up: All participants completed seven modules of treatment over twelve sessions, ten of which were 1:1 with the therapist and adolescent, and two of which also included the parent. Two additional optional parent-only sessions were offered as well. For each 1:1 session the parent was included for approximately ten minutes, generally at the end of the session, to discuss progress, the course of intervention content, and how the parent could assist with any take-home practice.
  Modules were adapted from the PI's intervention designed for ADHD in adults. Modules included: psychoeducation and organization/planning (4 session); distractibility (2 sessions); adaptive thinking/cognitive restructuring (2 sessions); procrastination (1 session); parent-adolescent sessions (2 sessions); parent-only sessions (1 session); relapse prevention (1 session).
- Wait List First, Then CBT: Participants initially assigned to the wait list were informed by the research assistant that they had been randomized to the wait list condition. For those who were still willing to cross-over to receive CBT, the research assistant contacted parents to schedule the 4-month assessment visit with the independent evaluator and the first CBT session after the evaluation for participants.
- Total: Total of all reporting groups
Arm/Group | CBT First, Then Follow-up | Wait List First, Then CBT | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.17 (1.01) | 15.09 (1.11) | 15.13 (1.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Changes in Attention Deficit Hyperactivity Disorder (ADHD) Symptoms - Adolescent Report
Description: -Independent blinded evaluator rated adolescent report of symptom severity (Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale-IV). The independent evaluator administered the ADHD rating scale-IV to adolescent participants. This scale, updated for Diagnostic and Statistical Manual of Mental Disorders, 4th Ed. (DSM-IV), assesses each of 18 individual symptoms of ADHD using an identical four-point severity grid (0 = not present up to 3 = severe; minimum total score = 0, maximum total score =54, with higher scores indicating greater symptomatology). The CBT for ADHD change score was calculated by combining the data for all participants who received CBT for ADHD (both those who received it between baseline and the 4-month assessment and those who received it between the 4-month and the 8-month assessment). The wait list control score represents only those participants who were in the wait list condition between the baseline and the 4-month assessment points.
Time Frame: before randomization, 4-months, 8-months
Population: The CBT group is comprised of participants originally randomized to receive CBT who completed the intervention (N=21) plus participants initially randomized to the wait-list group who crossed-over to receive CBT and completed the intervention (N=15). The wait list control group is comprised only of those initially assigned to the wait list (N=22).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Cognitive Behavioral Therapy (CBT) for ADHD: All participants completed seven modules of treatment over twelve sessions, ten of which were 1:1 with the therapist and adolescent, and two of which also included the parent. Two additional optional parent-only sessions were offered as well. For each 1:1 session the parent was included for approximately ten minutes, generally at the end of the session, to discuss progress, the course of intervention content, and how the parent could assist with any take-home practice.
  Modules were adapted from the PI's intervention designed for ADHD in adults. Modules included: psychoeducation and organization/planning (4 session); distractibility (2 sessions); adaptive thinking/cognitive restructuring (2 sessions); procrastination (1 session); parent-adolescent sessions (2 sessions); parent-only sessions (1 session); relapse prevention (1 session).
- Wait List Control: Participants initially assigned to the wait list were informed by the research assistant that they had been randomized to the wait list condition. For those who were still willing to cross-over to receive CBT, the research assistant contacted parents to schedule the 4-month assessment visit with the independent evaluator and the first CBT session after the evaluation for participants.
Arm/Group | Cognitive Behavioral Therapy (CBT) for ADHD | Wait List Control
Number analyzed (Participants) | 36 | 22
units on a scale | -4.27 (6.27) | -0.55 (5.72)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy (CBT) for ADHD vs Wait List Control; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; A longitudinal general linear mixed effects model was used; Mean Difference (Final Values) = 5.24, 95% CI 2-sided [3.28 to 7.21]

2. Primary Outcome: Attention Deficit Hyperactivity Disorder (ADHD) Symptom Severity - Clinician Rating
Description: -Independent, blinded evaluator rating of ADHD symptom severity (Clinical Global Impressions - severity scale). The Clinical Global Impression (CGI) Scale is a widely used rating scale to measure overall severity related to ADHD symptoms. The Global Severity rating ranges from; 1=not ill, to 7= extremely ill, with higher scores indicating greater severity.The CBT for ADHD change score was calculated by combining the data for all participants who received CBT for ADHD (both those who received it between baseline and the 4-month assessment and those who received it between the 4-month and the 8-month assessment). The wait list control score represents only those participants who were in the wait list condition between the baseline and the 4-month assessment points.
Time Frame: before randomization, 4-months, 8-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy (CBT) for ADHD | Wait List Control
Number analyzed (Participants) | 36 | 22
units on a scale | -1.14 (.83) | -0.09 (0.68)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy (CBT) for ADHD vs Wait List Control; Test type: Superiority or Other; p < .0001, Mixed Models Analysis; A longitudinal general linear mixed effects model was used; Mean Difference (Final Values) = 1.17, 95% CI 2-sided [.94 to 1.39]

3. Primary Outcome: Changes in Attention Deficit Hyperactivity Disorder (ADHD) Symptoms - Parent Report
Description: -Independent blinded evaluator rated parent report of symptom severity (ADHD Rating Scale-IV) to the parent of the adolescent participant. This scale, updated for Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV), assesses each of 18 individual symptoms of ADHD using an identical four-point severity grid (0 = not present up to 3 = severe; minimum total score = 0, maximum total score =54, with higher scores indicating greater symptomatology). The CBT for ADHD change score was calculated by combining the data for all participants who received CBT for ADHD (both those who received it between baseline and the 4-month assessment and those who received it between the 4-month and the 8-month assessment). The wait list control score represents only those participants who were in the wait list condition between the baseline and the 4-month assessment points.
Time Frame: baseline, 4-months, and 8-months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Behavioral Therapy (CBT) for ADHD | Wait List Control
Number analyzed (Participants) | 36 | 22
units on a scale | -9.27 (6.39) | -3.86 (6.84)
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy (CBT) for ADHD vs Wait List Control; Test type: Superiority; p < .0001, Mixed Models Analysis; A longitudinal general linear mixed effects model was used; Mean Difference (Net) = 10.93, 95% CI 2-sided [8.93 to 12.93]

ADVERSE EVENTS:
Time Frame: 8 months
Groups:
- CBT for ADHD First, Then Follow-up: All participants completed seven modules of treatment over twelve sessions, ten of which were 1:1 with the therapist and adolescent, and two of which also included the parent. Two additional optional parent-only sessions were offered as well. For each 1:1 session the parent was included for approximately ten minutes, generally at the end of the session, to discuss progress, the course of intervention content, and how the parent could assist with any take-home practice.
  Modules were adapted from the PI's intervention designed for ADHD in adults. Modules included: psychoeducation and organization/planning (4 session); distractibility (2 sessions); adaptive thinking/cognitive restructuring (2 sessions); procrastination (1 session); parent-adolescent sessions (2 sessions); parent-only sessions (1 session); relapse prevention (1 session).
- Wait List First, Then CBT for ADHD: Participants initially assigned to the wait list were informed by the research assistant that they had been randomized to the wait list condition. For those who were still willing to cross-over to receive CBT, the research assistant contacted parents to schedule the 4-month assessment visit with the independent evaluator and the first CBT session after the evaluation for participants.
Arm/Group | CBT for ADHD First, Then Follow-up | Wait List First, Then CBT for ADHD
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 0/24 | 0/22

LIMITATIONS AND CAVEATS:
* Initial efficacy trial leading to small sample size
* Sample was restricted to stably medicated adolescents
* Did not use a time-matched, attention-matched control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No